CLINICAL TRIAL: NCT05560958
Title: Post-market Clinical Follow-up Data Collection From Procedures With BIOTRONIK EP Products
Acronym: BIO|COLLECT-EP
Status: Recruiting | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: EP035
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BIOTRONIK EP catheters (AlCath, MultiCath, ViaCath), external devices (Qubic RF, Qubic Stim, Qiona) and transseptal sheaths (Senovo bi-flex) — Ablations and diagnostic catheters are indicated for temporary transvenous application in patients with cardiac arrhythmias during electrophysiology study (EPS) or catheter ablation interventions. They will be used in combination with external devices like RF generators, external pacemakers cardiac stimulators and / or irrigation pumps.

SUMMARY:
This data collection is designed to provide evidence for the safety, performance, and clinical benefit of BIOTRONIK's EP products. Additionally, residual risks will be monitored and newly emerging risks identified.

DETAILED DESCRIPTION:
In this study, data from routine care will be collected and evaluated to support regulatory post-market clinical follow-up demands under MDR as well as maintenance of the regulatory approval of the BIOTRONIK's EP product portfolio in the CE region. This is a prospective, observational, multi-center, international, open-label, non-randomized study that aims to provide evidence for the clinical safety, performance, and clinical benefit of BIOTRONIK's EP products. The patients participating in the study either receive a diagnostic or therapeutic catheter intervention, which are indicated for temporary transvenous application in patients with cardiac arrhythmias. They will be used in combination with external devices like RF generators, external pacemakers cardiac stimulators and / or irrigation pumps.

ELIGIBILITY:
Inclusion Criteria:

* Indication for diagnostic or therapeutic EP intervention
* EP intervention is planned to involve the use of BIOTRONIK EP products from at least 2 of the 3 following categories:

  * BIOTRONIK catheter (AlCath, ViaCath, MultiCath, Khelix)
  * BIOTRONIK external device (Qubic Stim, Qubic RF, Qiona)
  * BIOTRONIK transseptal sheath (Senovo Bi-Flex)
* BIOTRONIK EP product is planned to be used within its intended purpose
* Ability to understand the nature of the study
* Willingness to provide written informed consent
* Ability and willingness to perform all follow-up visits at the study site

Exclusion Criteria:

* Age less than 18 years
* Pregnant or breastfeeding
* Prior participation in this study with performed EP procedure
* Participation in an interventional clinical investigation in parallel to the BIO|COLLECT.EP study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for diagnosis and treatment of intracardiac arrhythmias in an EP lab environment.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Device deficiencies | During EP procedure
  Device deficiencies for each investigational device type that occur during the EP procedures in patients, users or other persons
Rate of Peri-procedural adverse device effects for each investigational device type | Until or at 24-hour follow-up
  Peri-procedural adverse device effects for each investigational device type that occur in all patients until or at the 24-hour follow-up
Rate of Post-procedural adverse device effects | After the 24-hour follow-up until or at the 3- to 6-month follow-up
  Post-procedural adverse device effects that occur in the AlCath group after the 24-hour follow-up until or at the 3- to 6-month follow-up
Percentage of Clinical benefit confirmations per number of use cases | At the time of procedure
  Clinical benefit at the time of procedure for each investigational device type

OTHER OUTCOMES:
Procedure setting (related to used BIOTRONIK EP products and competitor products) | Intervention
  Type of procedure, type of catheter models, recording system, RF ablation generator, irrigation pump, stimulator, 3D system, patient cable
Procedural parameters | Intervention
  Fluoroscopy time, Procedure duration, duration of RF energy delivery, date and time of procedure
Patient details | Baseline
  demographics, medical history, and concomitant cardiovascular medication
Device performance | Intervention
  e.g., successful insertion and advancing of catheter, successful stimulation and recording of intracardiac signals, RF energy application, removal, replacement/substitution of catheter, device used within its intended purpose

CONTACTS AND LOCATIONS:
Locations (1):
- Städtisches Krankenhaus Friedrichshafen, Friedrichshafen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Upon resonable request by authors or other scientifc reasons, but requires explicit approval by the sponsor.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available with uploading the results to clinical trial.gov. The data will be available as long as the study documents are archived.
Access Criteria: On demand; in case of request by an author or in case of scientific reasons, but requires explicit approval by the sponsor.